CLINICAL TRIAL: NCT01648712
Title: Platelet Function With New Pediatric Oxygenator and Heparin and Non Heparin Coating in Pediatric Cardiac Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: for difficulty to enroll patients in the study
Sponsor: Hôpital Necker-Enfants Malades (Other)
Collaborators: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Chiara Giorni, Doctor in Medicine, Hôpital Necker-Enfants Malades
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Necker
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Acquired Platelet Function Disorder
Keywords: extracorporeal circuit, platelet function
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Balance Circuit (Other): 24 patients will be assigned to the Balance group , using a non -heparin extracorporeal pediatric device for operation . The intervention is to use the Balance circuit for this arm
  Interventions: Device: non -heparin extracorporeal pediatric device for operation
- Carmeda Circuit (Other): 24 patients will be assigned to the Carmeda group, using a coated heparin extracorporeal pediatric device for operation.
  The intervention is to use the Carmeda circuit for this arm. The intervention is the Carmeda circuit.
  Interventions: Device: Balance surface, Carmeda heparin-coated surface

INTERVENTIONS:
Device: Balance surface, Carmeda heparin-coated surface — This study compares the influence of a Balance - coated CPB system in pediatric use versus the Carmeda TM heparin-coated system in platelet function preservation and hemostatic activation.
  Balance arm group recieved like intervention a Balance circuit
  Arms: Carmeda Circuit
Device: non -heparin extracorporeal pediatric device for operation — The carmeda arm group received like intervention the Carmeda circuit
  Arms: Balance Circuit

SUMMARY:
Optimal anticoagulation is mandatory during CPB in order to avoid hemostatic system activation. Platelet dysfunction is commonly observed after procedures performed under cardiopulmonary bypass (CPB). This is associated with a major risk of thrombosis and bleeding in the postoperative period.

Coating of the surface has been shown to diminish these effects.Biocompatible surfaces, extracorporeal circulation technologies mimic critical characteristics of the vascular endothelium to provide thromboresistance and enhanced blood compatibility. Recently, a new physiologic non heparin coating with different functional aspects was developed as an alternative to heparin based biological coatings. This bio-passive Hydrophilic Polymer Coating Without Heparin (BalanceTM Bio-Passive surface) and pediatric oxygenation system (Affinity PixieTM Oxygenation System), is designed to mimic the natural interfaces of blood. The aim of this study is to compare the influence of a Balance - coated CPB system in pediatric use versus the Carmeda TM heparin-coated system in platelet function preservation and hemostatic activation.

DETAILED DESCRIPTION:
Platelet dysfunction is commonly observed after procedures performed under cardiopulmonary bypass (CPB). This is associated with a major risk of thrombosis and bleeding in the postoperative period.

Coating of the surface has been shown to diminish these effects. Since the coagulation system and platelets are involved in the blood activation process, a coating might be a valuable approach to inhibit the different reactions. Improving the biocompatibility of the system by reduction of contact activation of blood elements is of significant importance, especially for neonates and infants who are more susceptible to the deleterious effects of extracorporeal circulation (ECC). Biocompatible surfaces extracorporeal circulation technologies mimic critical characteristics of the vascular endothelium to provide thromboresistance and enhanced blood compatibility. These biocompatible surfaces mitigate the foreign body response that occurs when blood comes in contact with non- endothelial surfaces.

Recently, a new physiologic non heparin coating with different functional aspects was developed as an alternative to heparin based biological coatings. This bio-passive Hydrophilic Polymer Coating Without Heparin (BalanceTM Bio-Passive surface) and pediatric oxygenation system (Affinity PixieTM Oxygenation System), is designed to mimic the natural interfaces of blood.

ELIGIBILITY:
Inclusion Criteria:

* Infants/children (weighting less than 18 Kg) undergoing surgical repair of congenital heart defects on CPB, presenting a saturation > 85% preoperatively.

Exclusion Criteria:

* Newborns, infants/children with Down syndrome, other syndromes or chromosomal abnormalities prematurity,
* use of circulatory arrest,
* expected perfusion time < 1 hour, documented coagulation disorders, use of anticoagulant or antiplatelet drugs within 48 hours of surgery, previous heart surgery and procedures requiring a return on CPB (2 or more CPB runs),
* cyanosis defined as oxygen saturation lower than 85%.

Ages: 30 Days to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the difference in levels of ß thromboglobulin (ß TG) at T2 (15 min after end of bypass) between the two groups. | six months
  Assuming a reduction of 30% of ß TG in infants treated with Balance TM , a total of 64 infants, 32 on each arm, will be needed to detect a Δ = 246 (mean ß TG = 820ng/ml in group Carmeda and mean ß TG =574ng/ml in group Balance; standard deviation=300) , in the level of ß TG at T2 with a two sided p=0.05 and a power of 80%.
  Taking in to account the use of non parametric test, we estimated an increase of the calculated sample size of 15%, yielding a total sample size of 74 patients.

SECONDARY OUTCOMES:
Platelet mapping by thromboelastography (Hemoscope, Medtronic) will be performed at the following times: T0,T1,T2,T3. | six months
  Flow cytometry will be analysed at T0, T1,T2. Fibrinogen levels, platelet count, prothrombin time, thrombin-antithrombin complex (TAT), F 1+2, PF4 , will be analysed at each time of the study.
  Differences of bleeding, and transfusion of any blood product, during the first postoperative 24 hours, will be collected.
  Analysis of differences of activation at different times, for two different temperatures, used for CPB in the two centers.
  Need of surgical review for bleeding, time of intubation, length of stay in ICU will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Giorni, M.D., Principal Investigator — Hopital Necker Enfants Malades
Locations (1):
- Hopital Necker Enfants Malades, Paris, France